CLINICAL TRIAL: NCT06072157
Title: A Phase 1, Double-Blind, Randomized, Placebo-Controlled, Sequential, Single- and Multiple-Ascending Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Immunogenicity of AK006 in Healthy Subjects and in Subjects With H1 Antihistamine Refractory Chronic Spontaneous Urticaria
Brief Title: Study to Assess the Safety, Tolerability, Pharmacokinetics and Immunogenicity of AK006 in Healthy Subjects and Subjects With Chronic Spontaneous Urticaria
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Allakos Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: AK006-001
Record Dates: First submitted 2023-09-09; First posted 2023-10-10 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-06

CONDITIONS: Healthy Participants; Chronic Spontaneous Urticaria
MeSH Terms: conditions — Chronic Urticaria

STUDY DESIGN:
Intervention Model Description: Single (Part A) and multiple (Part B) ascending IV dose study in healthy participants with a multiple dose expansion (Part C) in participants with chronic spontaneous urticaria. Single ascending (Part D) subcutaneous (SC) dose study in healthy participants
Who Masked: Participant, Investigator
Masking Description: Double-blind (placebo) essentially identical in appearance to the investigational drug (AK006)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Part A - Single Ascending Dose (SAD) Intravenous Cohorts (Experimental): Part A: Healthy adult participants will receive a single intravenous infusion of AK006 or matching placebo. The dose of AK006 will be increased per cohort. There will be up to 5 cohorts evaluated.
  Interventions: Drug: AK006-IV; Drug: Placebo-IV
- Part B - Multiple Ascending Dose (MAD) Intravenous Cohorts (Experimental): Part B: Healthy adult participants will receive multiple intravenous infusions of AK006 or matching placebo. The dose of AK006 will be increased per cohort. There will be up to 3 cohorts evaluated.
  Interventions: Drug: AK006-IV; Drug: Placebo-IV
- Part C - Multiple Dose Intravenous Cohort (Experimental): Part C: Adults with Chronic Spontaneous Urticaria will receive multiple intravenous infusions of AK006 or matching placebo.
  Interventions: Drug: AK006-IV; Drug: Placebo-IV
- Part D - Single Ascending Dose (SAD) Subcutaneous Cohorts (Experimental): Part D: Healthy adult participants will receive a single subcutaneous injection of AK006 or matching placebo. The dose of AK006 will be increased per cohort. There will be up to 2 cohorts evaluated.
  Interventions: Drug: AK006-SC; Drug: Placebo-SC

INTERVENTIONS:
Drug: AK006-IV — Intravenous infusion
  Arms: Part A - Single Ascending Dose (SAD) Intravenous Cohorts; Part B - Multiple Ascending Dose (MAD) Intravenous Cohorts; Part C - Multiple Dose Intravenous Cohort
Drug: Placebo-IV — Intravenous infusion
  Arms: Part A - Single Ascending Dose (SAD) Intravenous Cohorts; Part B - Multiple Ascending Dose (MAD) Intravenous Cohorts; Part C - Multiple Dose Intravenous Cohort
Drug: AK006-SC — Subcutaneous
  Arms: Part D - Single Ascending Dose (SAD) Subcutaneous Cohorts
Drug: Placebo-SC — Subcutaneous
  Arms: Part D - Single Ascending Dose (SAD) Subcutaneous Cohorts

SUMMARY:
This is a Phase 1, randomized, double-blind, placebo-controlled, sequential, single- and multiple-ascending dose study to evaluate the safety, tolerability, pharmacokinetics (PK), and immunogenicity of intravenous (IV) infusions and a single subcutaneous (SC) injection of AK006. The study will be conducted in 4 parts: a single-ascending dose part (Part A) in healthy participants, a multiple-ascending dose part (Part B) in healthy participants with an expanded cohort (Part C) in participants with chronic spontaneous urticaria (CSU), and a single ascending dose SC injection cohort (Part D) in healthy participants.

ELIGIBILITY:
Key Inclusion Criteria:

To be included in the study, the participant must:

* Weigh between 60 and 120 kg (inclusive) and have a body mass index (BMI) between 20 and 32 kg/m2, inclusive
* Agree (female of childbearing potential or male with female partner of childbearing potential) to use a highly effective method (<1% failure rate) of birth control, if sexually active from screening and for 16 weeks after the last dose of investigational product (IP).

Additionally, to be included in Part A, B and D, the participant must:

• Be in good general health with no significant medical history and has no clinically significant abnormalities on physical examination

Additionally, to be included in Part C, the participant must:

* Have a diagnosis of chronic spontaneous urticaria (CSU) for at least 6 months prior to screening
* Has a diagnosis of moderate to severe CSU that is refractory to stable doses of a single 2nd or later generation H1-AH between 1× and 4× the licensed dose and frequency at the time of randomization as defined by the following:

  * Presence of hives and itch for ≥6 consecutive weeks at any time prior to the Screening, despite the use of non-sedating H1-AHs. Note: Subject must be on a non-sedating H1-AH for treatment of CSU symptoms at the time of the Screening visit.
  * UAS7 score ≥16 with a HSS7 score ≥8 for the 2 consecutive weeks prior to randomization (Day 1) while on the stable dose of an H1-AH.
* Be on a stable dose of a single 2nd or later generation H1-antihistamines for the treatment of CSU, between 1× and 4× the licensed dose and frequency, by Day -14 of the Screening Period and must be willing to remain on the same stable dose throughout the study.
* Able and willing to complete a daily electronic diary to collect CSU symptoms for the duration of the study.

Key Exclusion Criteria:

A participant who meets any of the following exclusion criteria will not be eligible for inclusion in the study:

* Female participants who are pregnant, lactating, or planning to become pregnant during the study.
* Abnormal laboratory values, or findings in physical examination, ECG (QTc >450 ms for males and >470 ms for females), or vital signs considered to be clinically significant by the investigator.

Additionally, a participant will be excluded from Part A, B and D, if:

• Received treatment with any prescribed (excluding hormonal contraceptives or hormone replacement therapy [post-menopausal females]) or nonprescribed systemic or topical medication (including herbal product, and vitamins) within 21 days prior to the first dose of IP (excluding acetaminophen).

Additionally, a participant will be excluded from Part C, if:

* Has known or suspected urticarial vasculitis
* Subject has causes other than CSU for their urticaria including symptomatic dermographism, cholinergic urticaria, or any inducible urticaria
* Subject has other conditions or diseases that in the investigator's opinion might influence study evaluations and results
* Has any disease or condition (medical or surgical) which, in the opinion of the investigator, or medical monitor, would place the subject at increased risk

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-05-12 (Actual); Study Completion 2025-05-12 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events (AEs) | Screening to Day 113 (Part A and D), Screening to Day 141 (Part B), and Screening to Day 197 (Part C)
  AEs, serious AEs, and treatment emergent AEs (AE that starts after start of investigational product)
Incidence of AEs of special interest | Day 1 to Day 113 (Part A and D), Day 1 to Day 141 (Part B), and Day 1 to Day 197 (Part C)
  Infusion-related reactions, injection-related reactions, injection site reactions, anaphylaxis, and opportunistic infections
AEs leading to discontinuation | Day 1 to Day 113 (Part A and D), Day 1 to Day 141 (Part B), and Day 1 to Day 197 (Part C)
  AEs
Incidence of clinically significant abnormal laboratory values, electrocardiograms (ECGs), and vital signs | Day 1 to Day 113 (Part A and D), Day 1 to Day 141 (Part B), and Day 1 to Day 197 (Part C)
  Incidence of clinically significant abnormal laboratory values, electrocardiograms (ECGs), and vital signs

SECONDARY OUTCOMES:
AK006 serum concentration at end of IV infusion | Day 1 (Part A) and Day 29 (Part B)
  AK006 Serum concentration (ng/mL) at end of infusion
AK006 area under the concentration-time curve (AUC) from time 0 to the time of last quantifiable concentration (AUC[0-last]) | Day 1 to Day 113 (Part A and D) and Day 29 to Day 141 (Part B)
  AK006 AUC(0-last) (ng x h/mL)
AK006 AUC from time 0 extrapolated to infinity (AUC[0-inf]) | Day 1 to Day 113 (Part A and D)
  AK006 AUC(0-inf) (ng x h/mL)
Total systemic clearance of AK006 after intravenous or subcutaneous dose (CL) | Day 1 to Day 113 (Part A and D) and Day 1 to Day 141 (Part B)
  AK006 CL (L/h/kg)
Systemic steady-state volume of distribution (Vss) of AK006 | Day 1 to Day 113 (Part A and D) and Day 1 to Day 141 (Part B)
  AK006 Vss (mg/L)
AK006 Terminal elimination phase half-life (t1/2) | Day 1 to Day 113 (Part A and D) and Day 1 to Day 141 (Part B)
  AK006 t1/2 (hours)
Predose AK006 serum concentration (Ctrough, before the next dose) (Part B) | Day 29 (pre-dose)
  AK006 Ctrough (ng/mL)
AK006 AUC(0-last) after the second dose (Part B) | Day 29 to Day 141
  AK006 AUC(0-last) (ng x h/mL)
AK006 AUC over the dosing time interval (time 0 to 28 days) (AUC[tau]) (Part B) | Day 1 to Day 28 with each dosing interval
  AK006 AUC(tau) (ng x h/mL)
AK006 serum concentrations | Up to Day 141 (Part A, B, D); Up to Day 197 (Part C)
  AK006 ng/mL
AK006 absolute bioavailability subcutaneous injection | Day 1 to Day 113 (Part A and D)
  Ratio of mean AUC(0-last) after subcutaneous injection to mean AUC(0-last) after intravenous administration adjusted for dose
AK006 PK dose proportionality (Part A, B, D) | Up to Day 141
  Comparing dose-normalized Cmax and AUC (Part A, B, and D)
AK006 PK dose stationarity (Part B) | Up to Day 141
  Comparing AUCtau from last dose to AUCtau from first dose
AK006 Anti-drug Antibodies (ADAs) | Day 1 to Day 113 (Part A and D), Day 1 to Day 141 (Part B) and Day 1 to Day 197 (Part C)
  Number of participants with positive or negative AK006-ADAs

CONTACTS AND LOCATIONS:
Locations (25):
- United States (19):
  - Site 601-001 Healthy Volunteer Clinical Research Unit (Part A, B and D), Anniston, Alabama
  - Site 601-004 (Part C), Birmingham, Alabama
  - Site 601-008 (Part C), Scottsdale, Arizona
  - Site 601-014 (Part C), Bakersfield, California
  - Site 601-007 (Part C), Encino, California
  - Site 601-015 (Part C), Upland, California
  - Site 601-016 (Part C), Colorado Springs, Colorado
  - Site 601-006 (Part C), Overland Park, Kansas
  - Site 601-019 (Part C), Lexington, Kentucky
  - Site 601-003 (Part C), Baltimore, Maryland
  - Site 601-012 (Part C), Boston, Massachusetts
  - Site 601-023 (Part C), Troy, Michigan
  - Site 601-011 (Part C), St Louis, Missouri
  - Site 601-020 (Part C), Brooklyn, New York
  - Site 601-017 (Part C), Fargo, North Dakota
  - Site 601-002 (Part C), Cincinnati, Ohio
  - Site 601-018 (Part C), Portland, Oregon
  - Site 601-010 (Part C), El Paso, Texas
  - Site 601-013 (Part C), Greenfield, Wisconsin
- Canada (6):
  - Site 601-106 (Part C), Calgary, Alberta
  - Site 601-103 (Part C), London, Ontario
  - Site 601-107 (Part C), Niagara Falls, Ontario
  - Site 601-108 (Part C), Toronto, Ontario
  - Site 601-102 (Part C), Québec, Quebec
  - Site 601-105 (Part C), Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] O'Sullivan JA, Youngblood BA, Schleimer RP, Bochner BS. Siglecs as potential targets of therapy in human mast cell- and/or eosinophil-associated diseases. Semin Immunol. 2023 Sep;69:101799. doi: 10.1016/j.smim.2023.101799. Epub 2023 Jul 4. PMID 37413923